CLINICAL TRIAL: NCT03460990
Title: A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-659 Combination Therapy in Subjects With Cystic Fibrosis Who Are Homozygous for the F508del Mutation (F/F)
Brief Title: A Study of VX-659 Combination Therapy in CF Subjects Homozygous for F508del (F/F)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX17-659-103; 2017-004133-82 (EudraCT Number)
Record Dates: First submitted 2018-03-01; First posted 2018-03-09 (Actual); Results first posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor; tezacaftor, ivacaftor drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TEZ/IVA (Active Comparator): Following a run-in period of 4 weeks with Tezacaftor (TEZ)/Ivacaftor (IVA), participants received TEZ 100 milligram (mg)/IVA 150 mg as fixed-dose combination (FDC) tablet in the morning and IVA 150 mg as mono tablet in the evening for 4 weeks in the triple combination (TC) treatment period.
  Interventions: Drug: TEZ/IVA; Drug: IVA; Drug: Placebo
- VX-659/TEZ/IVA TC (Experimental): Following a run-in period of 4 weeks with TEZ/IVA, participants received VX-659 240 mg/TEZ 100 mg/IVA 150 mg as FDC tablets in the morning and IVA 150 mg as mono tablet in the evening for 4 weeks in the TC treatment period.
  Interventions: Drug: VX-659/TEZ/IVA; Drug: IVA; Drug: Placebo

INTERVENTIONS:
Drug: VX-659/TEZ/IVA — Participants received VX-659/TEZ/IVA orally once daily in the morning.
  Other Names: VX-659/VX-661/VX-770; VX-659/tezacaftor/ivacaftor
  Arms: VX-659/TEZ/IVA TC
Drug: TEZ/IVA — Participants received TEZ/IVA orally once daily in the morning.
  Other Names: VX-661/VX-770; tezacaftor/ivacaftor
  Arms: TEZ/IVA
Drug: IVA — Participants received IVA orally once daily in the evening.
  Other Names: VX-770; ivacaftor
Drug: Placebo — Participants received placebo matched TEZ/IVA orally once daily in the morning.
  Arms: VX-659/TEZ/IVA TC
Drug: Placebo — Participants received placebo matched to VX-659/TEZ/IVA orally once daily in the morning.
  Arms: TEZ/IVA

SUMMARY:
This study will evaluate the efficacy of VX-659 in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in subjects with cystic fibrosis (CF) who are homozygous for the F508del mutation (F/F).

ELIGIBILITY:
Key Inclusion Criteria:

* Homozygous for the F508del mutation (F/F)
* Forced expiratory volume in 1 second (FEV1) value ≥40% and ≤90% of predicted mean for age, sex, and height

Key Exclusion Criteria:

* Clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Solid organ or hematological transplantation

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Yale New Haven Medical Center, New Haven, Connecticut
  - University of Miami/Miller School of Medicine, Miami, Florida
  - St. Luke's CF Center of Idaho, Boise, Idaho
  - Advocate Children's Hospital- Park Ridge/ North Suburban Pulmonary and Critical Care Consultants, Niles, Illinois
  - Indiana Clinical Research Center, IU Health University Hospital, Indianapolis, Indiana
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Helen DeVos Children's Hospital CF Center, Grand Rapids, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine / St. Louis Children's Hospital, St Louis, Missouri
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Albany Medical College, Albany, New York
  - Northwell Health, Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Respiratory Diseases of Children and Adolescents, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sanford Research/ USD, Sioux Falls, South Dakota
  - University of Tennessee Medical Center-Adult Cystic Fibrosis Clinic, Knoxville, Tennessee
  - Children's Foundation Research Center/ Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah/ Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Australia (5):
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Adelaide Hospital, Adelaide
  - Prince Charles Hospital, Chermside
  - Institute for Respiratory Health Inc./ Sir Charles Gairdner Hospital, Nedlands
  - John Hunter Hospital & Hunter Medical Research Institute, New Lambton Heights
- Germany (2):
  - Charite Paediatric Pulmonology Department, Berlin
  - Pneumologische Praxis Pasing, München
- Ireland (3):
  - Cork University Hospital, Dublin
  - Our Lady's Children's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
- Spain (3):
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Universitari Vall d'Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (5):
  - Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridge
  - Liverpool Heart and Chest Hospital, Liverpool
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - University Hospital Llandough, Penarth

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 116 participants were enrolled in the study, of which 5 participants were included in the run-in period but were not dosed in TC treatment period. Results are presented for 111 participants dosed in the TC treatment period.
Pre-assignment Details: This study was conducted in participants with cystic fibrosis (CF) aged 12 years or older.
Period: Overall Study
Arm/Group | TEZ/IVA | VX-659/TEZ/IVA TC
Started | 57 | 54
Completed | 57 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TEZ/IVA: Following a run-in period of 4 weeks with TEZ/IVA, participants received TEZ 100 mg/IVA 150 mg as FDC tablet in the morning and IVA 150 mg as mono tablet in the evening for 4 weeks in the TC treatment period.
- Total: Total of all reporting groups
Arm/Group | TEZ/IVA | VX-659/TEZ/IVA TC | Total
Number analyzed (Participants) | 57 | 54 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (9.1) | 28.3 (9.6) | 27.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 26 | 59
  Male | 24 | 28 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 56 | 52 | 108
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 56 | 54 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Forced Expiratory Volume in 1 Second (ppFEV1) [Mean (Standard Deviation); unit: percentage points] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
  percentage points | 62.9 (14.9) | 62.0 (14.8) | 62.4 (14.8)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline at Week 4
Population: Full analysis set (FAS) included all randomized participants who carried the intended CF transmembrane conductance regulator gene (CFTR) allele mutation and received at least 1 dose of study drug in the TC Treatment Period.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Arm/Group | TEZ/IVA | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 57 | 54
percentage points | 0.3 (0.9) | 10.2 (0.9)
Statistical Analysis 1: Comparison: TEZ/IVA vs VX-659/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; Least Squares (LS) Mean Difference = 10, 95% CI 2-sided [7.4 to 12.5]

2. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline at Week 4
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | TEZ/IVA | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 57 | 54
millimole per liter (mmol/L) | 1.5 (1.8) | -47.2 (1.9)
Statistical Analysis 1: Comparison: TEZ/IVA vs VX-659/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = -48.7, 95% CI 2-sided [-53.9 to -43.5]

3. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline at Week 4
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEZ/IVA | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 57 | 54
units on a scale | 3.0 (1.7) | 16.5 (1.7)
Statistical Analysis 1: Comparison: TEZ/IVA vs VX-659/TEZ/IVA TC; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = 13.5, 95% CI 2-sided [8.8 to 18.3]

4. Secondary Outcome: Safety and Tolerability as Assessed Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug or to the completion of study participation date, whichever occurs first (up to Week 8)
Population: Safety set included all participants who received at least 1 dose of study drug in the TC treatment period.
Measure: Number; unit: participants
Arm/Group | TEZ/IVA | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 57 | 54
participants
  Participants with AEs | 31 | 33
  Participants with SAEs | 0 | 2

5. Secondary Outcome: Observed Pre-Dose Concentration (Ctrough) of VX-659, TEZ, TEZ Metabolite (M1-TEZ), and IVA
Time Frame: From Day 1 and Week 4
Population: Pharmacokinetic analysis set included all participants who received at least 1 dose of study drug in the TC treatment period. Here "Number analyzed" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | TEZ/IVA | VX-659/TEZ/IVA TC
Number analyzed (Participants) | 57 | 54
nanogram per milliliter (ng/mL)
  Day 1: VX-659: number analyzed (Participants) | 0 | 0
  Week 4: VX-659: number analyzed (Participants) | 0 | 52
  Week 4: VX-659 |  | 720 (589)
  Day 1: TEZ | 1780 (832) | 1590 (1020)
  Week 4: TEZ: number analyzed (Participants) | 56 | 53
  Week 4: TEZ | 1730 (885) | 1280 (594)
  Day 1: M1-TEZ | 5170 (1620) | 4840 (1860)
  Week 4: M1-TEZ: number analyzed (Participants) | 56 | 53
  Week 4: M1-TEZ | 5010 (1810) | 4730 (1380)
  Day 1: IVA | 717 (616) | 563 (400)
  Week 4: IVA: number analyzed (Participants) | 56 | 53
  Week 4: IVA | 722 (642) | 401 (211)

ADVERSE EVENTS:
Time Frame: From first dose of study drug in TC treatment period up to 28 days after last dose of study drug or to the completion of study participation date, whichever occurs first (up to Week 8)
Arm/Group | TEZ/IVA | VX-659/TEZ/IVA TC
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/57 | 2/54
Other Adverse Events (participants affected / at risk) | 19/57 | 23/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEZ/IVA (N=57) | VX-659/TEZ/IVA TC (N=54)
Depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TEZ/IVA (N=57) | VX-659/TEZ/IVA TC (N=54)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Alanine aminotransferase increased (Investigations) | 2 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 3
C-reactive protein increased (Investigations) | 0 | 4
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 9 | 2
Headache (Nervous system disorders) | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT03460990/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT03460990/SAP_001.pdf